Document: TDOC-0056233 Version: 1.0; CURRENT; Most-Recent; Effective

Status: Effective 

Title

# Clinical Evaluation of a Daily Wear Frequent Replacement Silicone Hydrogel Lens

Protocol Number: CLL949-C009 / NCT03920280

Development Stage of

Project:

Sponsor Name and Alcon Research, LLC. and its affiliates ("Alcon")

Address: 6201 South Freeway

Fort Worth, Texas 76134-2099

Test Product: LID015385

Property of Alcon
Confidential
May not be used, divulged, published, or otherwise disclosed without the consent of
Alcon


Status: Effective 

#### Investigator Agreement:

- I have read the clinical study described herein, recognize its confidentiality, and agree to conduct the described trial in compliance with Good Clinical Practice (GCP), the ethical principles contained within the Declaration of Helsinki, this protocol, all applicable regulatory authority regulations, and conditions of approval imposed by the reviewing IRB or regulatory authority.
- I will supervise all testing of the device involving human subjects and ensure that the requirements relating to obtaining informed consent and IRB review and approval are met in accordance with applicable local and governmental regulations.
- I have read and understand the appropriate use of the investigational product(s) as described in the protocol, current Investigator's Brochure, product information, or other sources provided by the Sponsor.
- I understand the potential risks and side effects of the investigational product(s).
- I agree to maintain adequate and accurate records in accordance with government regulations and to make those records available for inspection.
- I agree to comply with all other requirements regarding the obligations of clinical Investigators and all other pertinent requirements of the Sponsor and government agencies.
- I agree to ensure that all associates, colleagues, and employees assisting in the conduct of the study are informed of their obligations in meeting the above commitments.

| Have you ever been disqualified as an Investigator by any Regulatory Authority? | | |
|---|---|---|
| □ No □Yes | | |
| Have you ever been | involved in a study or other res | earch that was terminated? |
| □ No □Yes | | |
| If yes, please explai | n here: | |
| Principal Investigator: | | |
| | Signature | Date |
| Name and professional position: | | |
| Address: | | |


Status: Effective 

# **Table of Contents**

| Cl | inical Eva | aluation of a Daily Wear Frequent Replacement Silicone Hydrogel Lens | 1 |
|---|---|---|---|
| Ta | ble of Co | ntents | 3 |
| Lis | st of Table | es | 5 |
| Lis | st of Figu | res | 6 |
| 1 | GLOSS. | ARY OF TERMS | 7 |
| 2 | LIST O | F ACRONYMS AND ABBREVIATIONS | 11 |
| 3 | PROTO | COL SUMMARY | 13 |
| 5 | INTRO | DUCTION | 22 |
| | 5.1 | Rationale and Background | 22 |
| | 5.2 | Purpose of the Study | |
| | 5.3 | Risks and Benefits | 23 |
| 6 | STUDY | OBJECTIVES | 24 |
| | 6.1 | Primary Objective(s) | 24 |
| | 6.2 | Secondary Objective(s) | 24 |
| | 6.4 | Safety Objective(s) | 24 |
| 7 | INVEST | ΓΙGATIONAL PLAN | 25 |
| | 7.1 | Study Design | 25 |
| | 7.4 | Rationale for Choice of Control Product | 26 |
| | 7.5 | Data Monitoring Committee | 27 |
| 8 | STUDY | POPULATION | 27 |
| | 8.1 | Inclusion Criteria | 27 |
| | 8.2 | Exclusion Criteria | 28 |
| | 8.3 | Rescreening of Subjects | 29 |
| 9 | TREAT | MENTS ADMINISTERED | 29 |
| | 9.1 | Investigational Product(s) | 29 |


| Sta | tus: Effect | tive | |
|---|---|---|---|
| | 9.3 | Treatment Assignment / Randomization | 35 |
| | 9.4 | Treatment masking | 35 |
| | 9.5 | Accountability Procedures | 37 |
| | 9.6 | Changes to concomitant medications, treatments/ procedures | 38 |
| 10 | STUDY | PROCEDURES AND ASSESSMENTS | 38 |
| | 10.1 | Informed Consent and Screening | 39 |
| | 10.2 | Description of Study Procedures and Assessments | 40 |
| | | 10.2.1 Demographics | 40 |
| | | 10.2.2 Medical History and Concomitant Medications | |
| | | 10.2.3 Investigational Product Compliance | 40 |
| | | 10.2.4 Adverse Event Collection: Safety Assessment | 40 |
| | | 10.2.5 Slit-Lamp Biomicroscopy: Safety Assessment | |
| | | 10.2.6 Device Deficiencies: Safety Assessment | 40 |
| | 10.5 | | |
| | 10.5 | Discontinued Subjects | |
| | | 10.5.1 Screen Failures | |
| | | 10.5.2 Discontinuations | |
| | | 10.5.3 Schedule of Procedures and Assessments for Subjects Disc<br>from Investigational Product | |
| | 10.6 | Clinical Study Termination | 43 |
| | | 10.6.1 Follow-up of subjects after study participation has ended | 44 |
| 11 | ADVER | SE EVENTS AND DEVICE DEFICIENCIES | 44 |
| | 11.1 | General Information | 44 |
| | 11.2 | Monitoring for AEs | 47 |
| | 11.3 | Procedures for Recording and Reporting | 47 |
| | 11.5 | Unmasking of the Study Treatment | 50 |
| | 11.6 | Follow-Up of Subjects with AEs | 50 |
| | 11.7 | Pregnancy in the Clinical Study | 50 |
| 12 | ANALY | SIS PLAN | 51 |
| | 12.1 | Subject Evaluability | 51 |
| | | Analysis Sets | 51 |

| Alcon - Bus<br>Document: TD | Version: 1.0; CURRENT; Most-Recent; Effective | <b>Date:</b> 22-Mar-2019 |
|---|---|---|
| Status: Effect | | |
| 12.3 | Demographic and Baseline Characteristics | 51 |
| 12.4 | Effectiveness Analyses | 51 |
| | 12.4.1 Analysis of Primary Effectiveness Endpoint(s) | 52 |
| | 12.4.1.1 Statistical Hypotheses | |
| | 12.4.1.2 Analysis Methods | 52 |
| 12.5 | Handling of Missing Data | 53 |
| 12.6 | Safety Analyses | 53 |
| 13 DATA H | ANDLING AND ADMINISTRATIVE REQUIREMENTS | 54 |
| 13.1 | Subject Confidentiality | 54 |
| 13.2 | Completion of Source Documents and Case Report Forms | 55 |
| 13.3 | Data Review and Clarifications | 56 |
| 13.4 | Sponsor and Monitoring Responsibilities | 56 |
| 13.5 | Regulatory Documentation and Records Retention | |
| 13.6 | Quality Assurance and Quality Control | 57 |
| 14 ETHICS | | 57 |
| 15 REFERI | ENCES | 58 |
| 15.1 | References applicable for all clinical studies | 58 |
| | 15.1.1 US references applicable for clinical studies | 58 |
| | List of Tables | |
| Table 2–1 | List of Acronyms and Abbreviations Used in This Protocol | 11 |
| Table 3–1 | Schedule of Study Procedures and Assessments | |
| | • | |
| Table 6–1 | Primary Objective(s) | |
| Table 6–2 | Safety Objective(s) | 24 |
| Table 9–1 | Test Product | 30 |

| -Mar-2019 |
|---------------------------|
| ge <b>6</b> of <b>5</b> 9 |
| 32 |
| 26 |
| 44 |
| 45 |


Status: Effective 

## 1 GLOSSARY OF TERMS

| Names of test product(s) | Throughout this document, test product(s) will be referred to |
|---|---|
| | as soft contact lenses |
| Name of Control Product(s) | CooperVision® BIOFINITY® soft contact lenses (Biofinity |
| | contact lenses or Biofinity) |
| Adverse Device Effect | Adverse event related to the use of an investigational |
| (ADE) | medical device (test product) or control product. Note: This |
| | definition includes adverse events resulting from insufficient |
| | or inadequate instructions for use, deployment, |
| | implantation, installation, or operation; any malfunction; |
| | and use error or intentional misuse of the test product or |
| | control product. |
| Adverse Event (AE) | Any untoward medical occurrence, unintended disease or |
| raverse Event (rie) | injury, or untoward clinical signs (including abnormal |
| | laboratory findings) in subjects, users or other persons, |
| | whether or not related to the investigational medical device |
| | (test product). Note: For subjects, this definition includes |
| | events related to the test product, the control product, or the |
| | procedures involved. For users or other persons, this |
| | definition is restricted to events related to the test product. |
| | Requirements for reporting Adverse Events in the study can |
| | be found in Section 11. |
| Anticipated Serious | Serious adverse device effect which by its nature, incidence, |
| Adverse Device Effect | severity, or outcome has been identified in the risk |
| | management file. |
| Device Deficiency | Inadequacy of a medical device with respect to its identity, |
| | quality, durability, reliability, safety, or performance. Note: |
| | This definition includes malfunctions, use errors, and |
| | inadequate labeling. |


Status: Effective 

| | Requirements for reporting Device Deficiencies in the study |
|---|---|
| | can be found in Section 11. |
| Enrolled Subject | Any subject who signs an informed consent form for |
| | participation in the study. |
| Interventional Clinical Trial | A research trial that prospectively assigns, whether |
| | randomly or not, human participants or groups of humans to |
| | one or more health-related interventions to evaluate the |
| | effects on health outcomes, and/or a research trial in which |
| | diagnostic or monitoring procedures beyond standard of care |
| | are conducted and generate outcomes for use in analysis of |
| | data. |
| I (: 4: 1D 1 4 | |
| Investigational Product | Is defined as a preventative (vaccine), a therapeutic (drug or |
| | biologic), device, diagnostic, or palliative used as a test or |
| | control product in a clinical trial, including a product with a |
| | marketing authorization when used or assembled |
| | (formulated or packaged) in a way different from the |
| | authorized form, or when used for an unauthorized |
| | indication, or when used to gain further information about |
| | the authorized form. |
| | the authorized form. |
| Malfunction | Failure of a medical device to perform in accordance with its |
| | intended purpose when used in accordance with the |
| | instructions for use or clinical investigation plan. |
| | instructions for use of crimear investigation plan. |
| Non-serious Adverse Event | Adverse event that does not meet the criteria for a serious |
| Tion serious ruverse Event | adverse event. |
| | adverse event. |
| Randomized Subjects | Any subject who is assigned a randomized treatment. |
| Tanaomizoa baojeoto | 2 mg 5 do good 11 no 15 do signed a randomized treatment. |
| Serious Adverse Device | Adverse device effect that has resulted in any of the |
| Effect (SADE) | consequences characteristic of a serious adverse event. |
| , , , | 1 |
| Serious Adverse Event | Adverse event that led to any of the following: |
| (SAE) | |
| | • Death. |


Status: Effective 

• A serious deterioration in the health of the subject that either resulted in:

- a. a life-threatening illness or injury.

  Note: Life-threatening means that the individual was at immediate risk of death from the event as it occurred, ie, it does not include an event which hypothetically might have caused death had it occurred in a more severe form.
- b. any potentially sight-threatening event or permanent impairment to a body structure or a body function.
- c. in-patient hospitalization or prolonged hospitalization.

Note: Planned hospitalization for a preexisting condition, without serious deterioration in health, is not considered a serious adverse event. In general, hospitalization signifies that the individual remained at the hospital or emergency ward for observation and/or treatment (usually involving an overnight stay) that would not have been appropriate in the physician's office or an out-patient setting. Complications that occur during hospitalization are adverse events. If a complication prolongs hospitalization or fulfills any other serious criteria, the event is serious. When in doubt as to whether "hospitalization" occurred, the event should be considered serious.

- d. a medical or surgical intervention to preventa) or b).
- e. any indirect harm as a consequence of incorrect diagnostic test results when used within manufacturer's instructions for use.


Status: Effective 

| | Fetal distress, fetal death, or a congenital abnormality or birth defect. Refer to Section 11 for additional SAEs. |
|---|---|
| Significant Non-Serious<br>Adverse Event | Is a symptomatic, device-related, non-sight threatening adverse event that warrants discontinuation of any contact lens wear for greater than or equal to 2 weeks. Refer to Section 11 for additional Significant Non-Serious AEs. |
| Unanticipated Serious<br>Adverse Device Effect | Serious adverse device effect which by its nature, incidence, severity or outcome has not been identified in the risk management file. |
| Use Error | Act or omission of an act that results in a different medical device response than intended by manufacturer or expected by user. Note: This definition includes slips, lapses, and mistakes. An unexpected physiological response of the subject does not in itself constitute a use error. |


Status: Effective 

### 2 LIST OF ACRONYMS AND ABBREVIATIONS

Table 2-1 List of Acronyms and Abbreviations Used in This Protocol

| Abbreviation | Definition |
|---|---|
| ADE | Adverse device effect |
| AE | Adverse event |
| BCVA | Best corrected visual acuity |
| Biofinity contact lens | CooperVision BIOFINITY (comfilcon A) soft contact lenses |
| or Biofinity | |
| CFR | Code of Federal Regulations |
| CLEAR CARE | CLEAR CARE Cleaning & Disinfecting Solution |
| CRF | Case report form |
| CSM | Clinical site manager |
| CTT | Clinical trial team |
| D | Diopter(s) |
| D/C | Discontinue |
| eCRF | Electronic case report form |
| EDC | Electronic data capture |
| FDA | US Food and Drug Administration |
| GCP | Good Clinical Practice |
| IB | Investigator's brochure |
| ICF | Informed consent form |
| ICH | International Council for Harmonisation of Technical |
| | Requirements for Pharmaceuticals for Human Use |
| IEC | Independent ethics committee |
| IP | Investigational product |
| IRB | Institutional review board |
| ISO | International Organization for Standardization |
| LID | Lens identification |
| logMAR | Logarithm of the minimum angle of resolution |
| mm | Millimeter |
| N/A | Not applicable |
| OD | Right eye |
| OS | Left eye |
| OU | Both eyes |
| SAE | Serious adverse event |


Status: Effective 

| Abbreviation | Definition |
|--------------|-------------------------------|
| SADE | Serious adverse device effect |
| SiHy | Silicone hydrogel |
| SOP | Standard operating procedure |
| US / USA | United States of America |
| USAN | United States Adopted Name |
| USV | Unscheduled visit |
| VA | Visual acuity |
| VS | Versus |


Status: Effective 

## 3 PROTOCOL SUMMARY

| This will be a prospective, randomized double-masked, parallel-group clinical study. | controlled, |
|---|---|
| Approximately 8 sites in the US will enroll approximately 120 subjects. Subjects expected to attend 6 office visits: Screening / Baseline / Dispense, Week 1 Fol Follow-up, Month 1 Follow-up, Month 2 Follow-up and Month 3 Follow up/Expected duration of participation for each subject is approximately 3 months wear clinical study. Approximately 80 subjects will be assigned to wear the testilization for each subjects will be assigned to wear the testilization of participation for each subjects will be assigned to wear the testilization of participation for each subjects will be assigned to wear the testilization for each subjects will be assigned to wear the testilization for each subjects will be assigned to wear the control lenses, | llow up, Week 2<br>Exit. The total<br>in this daily |
| Subjects and the study personnel conducting the study evaluations will be mast treatment. Subjects who meet the inclusion and exclusion criteria will be rand either the test contact lenses in both eyes or the control contact lense in both eyes for 3 months of daily wear exposure. | omized to wear |
| At the Screening / Baseline / Dispense Visit, study lenses will be dispensed to subjects | qualified |
| All study lenses will be worn for at least 5 days per week and 8 hours per day modality (eg, will not be worn while sleeping). | in a daily wear |
| Regardless of whether the subject is randomized to the test group, CLEAR CARE® Cleaning & Disinfecting Solution (CLEAR CARE) in | |
| cleaning and disinfection. | Tast oc asca for |


Status: Effective 

| <u>.</u> |
|----------|

| Investigational | Medical Device |
|---|---|
| Investigational | Medical Device |
| product type | |
| Study type | Interventional |
| Investigational | Test Product: soft contact lens |
| products | Control Product: Biofinity soft contact lens |
| Purpose and | The purpose of this clinical study is to demonstrate the |
| rationale | performance of the investigational soft contact lens |
| | compared to the commercially available Biofinity soft contact lens |
| | when worn in a daily wear modality, by assessing visual acuity as |
| | the primary variable. |
| Objective(s) | The primary objective is to demonstrate safety and effectiveness of |
| | the soft contact lens when worn for daily wear as |
| | compared to the Biofinity soft contact lens. |
| Endpoint(s) | Primary Effectiveness |
| | Distance VA (Snellen) |


Status: Effective 

| Status. ======= | 1 110 10 01 0 |
|-----------------|-----------------------------------------|
| | Safety |
| | • AEs |
| | Biomicroscopy findings |
| | Device deficiencies |
| Assessment(s) | Effectiveness |
| | VA with study lenses (Snellen distance) |
| | · <del></del> |
| | <u> </u> |


Status: Effective 

| Status: Effective | 1 age 10 01 37 |
|---|---|
| Study Design | Safety AEs Biomicroscopy Device deficiencies This will be a prospective, randomized, controlled, double-masked, parallel-group, daily |
| | wear clinical study. Subject participation in the study will be approximately 14 weeks with approximately 3 months of exposure to study lenses. |
| Subject population | Volunteer subjects aged 18 or over who are adapted daily wear frequent replacement soft contact lens wearers, excluding Biofinity habitual wearers, have at least 3 months of soft contact lens wearing experience, and who wear their habitual lenses at least 5 days per week and at least 8 hours per day. |
| Key inclusion criteria (See Section 8.1 for a | <ul> <li>Successful wear of spherical daily wear frequent<br/>replacement soft contact lenses for distance correction in<br/>both eyes during the past 3 months for a minimum of 5 days<br/>per week and 8 hours per day.</li> </ul> |


Status: Effective 

| _ | |
|---|---|
| complete list of inclusion criteria) | • Manifest cylinder ≤ 0.75 D in each eye |
| Key exclusion criteria (See Section 8.2 for a complete list of exclusion criteria) | <ul> <li>Wearing habitual contact lenses in an extended wear modality (routinely sleeping in lenses for at least 1 night per week) over the last 3 months prior to enrollment.</li> <li>Monovision contact lens wearers</li> <li>Habitually wearing Biofinity lenses</li> </ul> |
| Data analysis and sample size justification | effectiveness and safety data will be presented separately based |
| | upon subject study status of Completed or Discontinued. No formal hypotheses are formulated for the primary effectiveness endpoint, hence no inferential testing will be performed. |
| Key words | Biofinity, daily wear, |
| Associated materials | CLEAR CARE Cleaning & Disinfecting Solution will be used for daily cleaning and disinfection. |

Alcon - Business Use Only Protocol - Clinical Document: TDOC-0056233 Version: 1.0; CU Status: Effective

Table 3-1 Schedule of Study Procedures and Assessments

| Procedure/ Assessment | Visit 1 Screening/ Baseline/ Dispense | Visit 2<br>Week 1<br>Follow-up | Visit 3<br>Week 2<br>Follow-up | Visit 4 Month 1 Follow-up | Visit 5 Month 2 Follow-up | Visit 6 Month 3 Follow-up/Exit | Early<br>Exit | USV |
|---|---|---|---|---|---|---|---|---|
| | Day 1 | Day 7 | Day 15 | Day 30 | Day 60 | Day 95 | | |
| Informed Consent | ✓ | - | - | - | - | - | - | - |
| Demographics | ✓ | - | - | - | - | - | - | - |
| Medical History | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | (✓) |
| Concomitant Medications | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | (✓) |
| Inclusion/ Exclusion | ✓ | - | - | - | - | - | - | - |
| Habitual lens information<br>(brand / manufacturer,<br>modality, power, wear<br>success, habitual lens care<br>brand) | ✓ | - | - | - | - | - | - | - |
| | | I | I | I | I | | | |

| Procedure/ Assessment | Visit 1 Screening/ Baseline/ Dispense | Visit 2<br>Week 1<br>Follow-up | Visit 3<br>Week 2<br>Follow-up | Visit 4<br>Month 1<br>Follow-up | Visit 5 Month 2 Follow-up | Visit 6<br>Month 3<br>Follow-up/Exit | Early<br>Exit | USV |
|---|---|---|---|---|---|---|---|---|
| | Day 1 | Day 7 | Day 15 | Day 30 | Day 60 | Day 95 | | |
| Biomicroscopy | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | (✓) |
| | | I | I | I | I | I | ı | I |
| Randomize | ✓ | - | - | - | - | - | - | - |
| IP Dispense | ✓ | ✓ | (✔) | (✔) | (✓) | - | - | (✓) |
| VA w/ study lenses<br>(OD, OS Snellen distance) <sup>1</sup> | ✓ | ✓ | ✓ | ✓ | ✓ | <b>✓</b> | ✓ | (✓) |

Print Date:

| Status: Effective | Document: TDOC-0056233 | Alcon - Business Use Only Protocol - Clinical |
|---|---|---|
| | Version: 1.0; CURRENT; Most-Recent; Effective | otocol - Clinical |
| | t-Recent; Eff | |
| | fective | Effective Date: 3/22/2 |

| Procedure/ Assessment | Visit 1 Screening/ Baseline/ Dispense | Visit 2 Week 1 Follow-up | Visit 3 Week 2 Follow-up Day 15 | Visit 4 Month 1 Follow-up | Visit 5 Month 2 Follow-up Day 60 | Visit 6 Month 3 Follow-up/Exit Day 95 | Early<br>Exit | USV |
|---|---|---|---|---|---|---|---|---|
| | I | | | | | | | |
| | ı | | | | | | | |

Alcon - Business Use Only Protocol - Clinical Document: TDOC-0056233 Version: 1.0; CU Status: Effective

| Procedure/ Assessment | Visit 1 Screening/ Baseline/ Dispense | Visit 2<br>Week 1<br>Follow-up | Visit 3<br>Week 2<br>Follow-up | Visit 4 Month 1 Follow-up | Visit 5 Month 2 Follow-up | Visit 6 Month 3 Follow-up/Exit | Early<br>Exit | USV |
|---|---|---|---|---|---|---|---|---|
| | Day 1 | Day 7 | Day 15 | Day 30 | Day 60 | Day 95 | | |
| AEs | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | (✓) |
| Device deficiencies | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | (✔) |
| Exit Form | (✓) | (✓) | (✓) | (✓) | (✓) | ✓ | ✓ | (✓) |

a) All follow-up visits should be scheduled at least 4 hours after lens insertion

Effective Date: 22-Mar-2019




Status: Effective 



Refer to the IB for additional information.

### **6 STUDY OBJECTIVES**

## 6.1 Primary Objective(s)

Table 6–1 Primary Objective(s)

| Objective(s) | Endpoint(s) |
|---|---|
| Demonstrate safety and effectiveness of | Primary Effectiveness |
| soft contact lens when worn for daily wear as compared to Biofinity soft | • Distance VA (Snellen) |
| contact lens. | |

# 6.2 Secondary Objective(s)

Not Applicable



# 6.4 Safety Objective(s)

Table 6–2 Safety Objective(s)

| Objective(s) | Endpoint(s) |
|-----------------------------------------------|------------------------|
| Duty of care and evaluation of safety profile | AEs |
| of the investigational products. | Biomicroscopy findings |
| | Device deficiencies |


Status: Effective 

### 7 INVESTIGATIONAL PLAN

### 7.1 Study Design

| This will be a prospective, randomized, | controlled, |
|-----------------------------------------------------------|-------------|
| double-masked, parallel-group, daily wear clinical study. | |

This clinical study will engage approximately 8 clinic sites to enroll approximately 120 subjects with approximately 15 subjects per site.

Subjects will be expected to attend 6 office visits: Screening / Baseline / Dispense, Week 1 Follow-up, Week 2 Follow-up, Month 1 Follow-up, Month 2 Follow-up, and Month 3 Follow up/Exit. The total expected duration of participation for each subject is approximately 3 months in this daily wear study. Subjects will be randomized to wear either the test contact lenses in both eyes or the control Biofinity contact lenses in both eyes.

| Following randomization, study lenses will be dispensed to the subject. |
|---|
| Subjects will wear the lenses while awake in a daily wear modality. CLEAR CARE will be |
| used for daily cleaning and disinfection. |


Status: Effective 



Figure 7-1 Flowchart of Study Visits





#### 7.4 Rationale for Choice of Control Product




Status: Effective 

persons with non-diseased eyes.

### 7.5 Data Monitoring Committee

Not Applicable

#### 8 STUDY POPULATION

The study population consists of adult male or female subjects (aged 18 or over), with non-diseased eyes, who require optical correction for refractive ametropia.

The intended study population consists of volunteer subjects who are frequent replacement daily wear soft contact lens wearers, excluding Biofinity habitual wearers, who have at least 3 months of contact lens wearing experience, and who wear their habitual lenses at least 5 days per week and 8 hours per day.

#### 8.1 Inclusion Criteria

Written informed consent must be obtained before any study specific assessment is performed. Upon signing informed consent, the subject will be considered enrolled in the study.

Subjects eligible for inclusion in this study must fulfill all of the following criteria:

- At least 18 years of age and be able to understand and sign an IRB/IEC approved Informed Consent form.
- 2. Willing and able to attend all scheduled study visits as required per protocol.
- Successful wear of spherical daily wear frequent replacement soft contact lenses for distance correction in both eyes during the past 3 months for a minimum of 5 days per week and 8 hours per day.
- 4. Manifest cylinder  $\leq 0.75$  D in each eye.


Status: Effective 

## 8.2 Exclusion Criteria

Subjects fulfilling any of the following criteria are not eligible for participation in this study.



| Document: TDOC-0056233 Status: Effective | Version: 1.0; CURRENT; Most-Recent; Effective | Page <b>29</b> of <b>59</b> |
|---|---|---|
| | t lenses in an extended wear modality (routinely per week) over the last 3 months prior to enroll | |
| 13. Monovision wearers. | | |
| 16. Any habitual wear of Bio | ofinity lenses. | |
| Women of childbearing potentian not excluded from participation. | al or women who are pregnant at the time of stud | ly entry are |
| not excluded from participation. | | |
| 8.3 Rescreening of Subje | ects | |
| Rescreening of subjects is not al | llowed in this study. | |
| 9 TREATMENTS ADM | INISTERED | |
| 9.1 Investigational Prod | · · · <u> </u> | |
| Test Product(s): | soft contact lenses | |
| Control Product(s) | Biofinity (comfilcon A) soft contact lense | es . |

Effective Date: 22-Mar-2019

Printed By: Print Date:

 $Alcon \textbf{-} Business \ Use \ Only \ {\tt Protocol} \ \textbf{-} \ {\tt Clinical}$ 


Status: Effective 

Table 9–1 Test Product

| Test Product | soft contact lenses ( contact lens) |
|---|---|
| | (LID015385) |
| Manufacturer | Alcon Vision, LLC. 6201 South Freeway Fort Worth, Texas 76134-2099 USA |
| Indication for use and intended purpose in the current study | The intended use of this contact lens is for vision correction. |
| Product description<br>and parameters<br>available for this<br>study | |
| Usage | <ul> <li>Wear: <ul> <li>Daily Wear</li> <li>During waking hours only.</li> </ul> </li> <li>Bilateral</li> <li>Exposure: At least ~8 hours per day and ~5 days per week over a ~3 month exposure period.</li> </ul> |


Status: Effective 






Status: Effective 

**Table 9–2** Control Product

| Control Product(s) | Biofinity (comfilcon A) soft contact lenses (Biofinity contact lens) (LID010221) |
|---|---|
| Manufacturer | CooperVision |
| Indication for Use | The intended use of this contact lens is for vision correction. |
| Product description<br>and parameters<br>available for this<br>study | <ul> <li>Material: comfilcon A</li> <li>Water content: 48%</li> <li>Power range: -1.00 to -6.00 D (0.25 D steps)</li> <li>Base curve: 8.6 mm (target)</li> <li>Diameter: 14.0 mm (target)</li> </ul> |
| Formulation | Silicone Hydrogel. Additional details can be found in the Biofinity package insert. |
| Usage | Wear: O Daily Wear |


Status: Effective 



 $Alcon \textbf{-} Business \ Use \ Only \ \texttt{Protocol} \ \textbf{-} \ \texttt{Clinical}$ Effective Date: 22-Mar-2019

Version: 1.0; CURRENT; Most-Recent; Effective Document: TDOC-0056233

Status: Effective 



More information on the test product can be found in the IB; information on the control product can be found in the Package Insert.

| _ |
|---|




Status: Effective 
Effective Date: 22-Mar-2019 Alcon - Business Use Only Protocol - Clinical Version: 1.0; CURRENT; Most-Recent; Effective Document: TDOC-0056233 Status: Effective  **Accountability Procedures** 9.5

It is the Investigator's responsibility to ensure that:

- All study products are accounted for and not used in any unauthorized manner
- •


Status: Effective 

• All unused products are available for return to the Study Sponsor, as directed

Any study lenses associated with a device deficiency or with any product-related AE
(ie, ADE or SADE) are returned to the Study Sponsor for investigation, unless
otherwise directed by the Sponsor. Refer to Section 11 of this protocol for additional
information on the reporting of device deficiencies and AEs

The Investigator is responsible for proper disposition of all unused IPs at the conclusion of the study,

## 9.6 Changes to concomitant medications, treatments/ procedures

After the subject is enrolled into the study, the Investigator must instruct the subject to notify the study site about:

- Any new medications
- Alterations in dose or dose schedules for current medications,
- Any medical procedure or hospitalization that occurred or is planned
- Any non-drug therapies (including physical therapy and blood transfusions).

The Investigator must document this information in the subject's case history source documents.

#### 10 STUDY PROCEDURES AND ASSESSMENTS

Subjects will be expected to attend 6 office visits, as shown below.

| Visit # | Visit Type | Visit Day |
|---------|-------------------------------------------|-----------|
| Visit 1 | Screening/Baseline/Randomization/Dispense | Day 1 |
| Visit 2 | Week 1 Follow-up Visit | Day 7 |
| Visit 3 | Week 2 Follow-up Visit | Day 15 |
| Visit 4 | Month 1 Follow-up Visit | Day 30 |
| Visit 5 | Month 2 Follow-up Visit | Day 60 |
| Visit 6 | Month 3 Follow-up / Exit Visit | Day 95 |


Status: Effective 



At the Screening / Baseline / Dispense Visit, study lenses will be dispensed to the subject. All subjects will wear the study lenses in a daily wear modality, only during waking hours.



# 10.1 Informed Consent and Screening

The Investigator or delegate must explain the purpose and nature of the study, and have the subject read, sign, and date the IRB/IEC-approved informed consent document. The subject must sign the ICF BEFORE any study-specific procedures or assessments can be performed, including study-specific screening procedures. Additionally, have the individual obtaining consent from the subject and a witness, if applicable, sign and date the informed consent document.


Status: Effective 

The Investigator or delegate must provide a copy of the signed document to the subject and place the original signed document in the subject's chart, or provide documentation as required by local regulations.

## 10.2 Description of Study Procedures and Assessments

The

Investigator is responsible for ensuring responsibilities for all procedures and assessments are delegated to appropriately qualified site personnel.

## 10.2.1 Demographics

Obtain demographic information including age, race, ethnicity, and sex.

## 10.2.2 Medical History and Concomitant Medications

Collect medical history information, including information on all medications used within the past 30 days. Include herbal therapies, vitamins, and all over-the-counter as well as prescription medications. Throughout the subject's participation, obtain information on any changes in medical health and/or the use of concomitant medications.

# 10.2.3 Investigational Product Compliance

Review subject compliance with the study lenses usage and adjunct product usage

# 10.2.4 Adverse Event Collection: Safety Assessment

Assess and record any AEs that are observed or reported, including those associated with changes in concomitant medication dosing since the previous visit. Requirements for reporting AEs in the study can be found in Section 11.

# 10.2.5 Slit-Lamp Biomicroscopy: Safety Assessment

Slit-lamp examination of the cornea, iris/anterior chamber, and lens must be performed in both eyes before instillation of any diagnostic eye drops.

# 10.2.6 Device Deficiencies: Safety Assessment

Assess and record any device deficiencies that are reported or observed since the previous visit. Requirements for reporting device deficiencies in the study can be found in Section 11.


Status: Effective 



Document: TDOC-0056233

Version: 1.0; CURRENT; Most-Recent; Effective


Effective Date: 22-Mar-2019

# 10.5 Discontinued Subjects

Alcon - Business Use Only Protocol - Clinical

#### 10.5.1 Screen Failures

Screen failures are subjects who were excluded from the study after signing the informed consent, not meeting the inclusion/exclusion criteria, and prior to randomization to product/dispense of study product.

The Investigator must document the reason for screen failure in the subject's case history source documents.

Subject numbers must not be re-used.

#### 10.5.2 Discontinuations

Discontinued subjects are individuals who voluntarily withdraw or are withdrawn from the study by the Investigator after signing the informed consent.

Subject numbers of discontinued subjects must not be re-used.


Status: Effective 

Subjects may discontinue from study or study treatment at any time for any reason. Subjects may also be discontinued from study treatment at any time if, in the opinion of the Investigator, continued treatment poses a risk to their health.



## **10.6 Clinical Study Termination**

The Study Sponsor reserves the right to close the investigational site or terminate the study in its entirety at any time.

If the clinical study is prematurely terminated or suspended by the Study Sponsor:

- The Study Sponsor must:
  - o Immediately notify the Investigator(s) and subsequently provide instructions for study termination.
  - o Inform the Investigator and the regulatory authorities of the termination/suspension and the reason(s) for the termination/suspension.
- The Investigator must:
  - Promptly notify the IRB/IEC of the termination or suspension and of the reasons.
  - Provide subjects with recommendations for post-study treatment options as needed.


Status: Effective 

The Investigator may terminate the site's participation in the study for reasonable cause.

# 10.6.1 Follow-up of subjects after study participation has ended

Following this study, the subject will return to their eye care professional for their routine eye care.

#### 11 ADVERSE EVENTS AND DEVICE DEFICIENCIES

### 11.1 General Information

An AE is any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users, or other persons, whether or not related to the investigational medical device (test article). Refer to the Glossary of Terms and figures below for categories of AEs and SAEs.

Figure 11–1 Categorization of All AEs




Status: Effective 

Figure 11-2 Categorization of All SAE



#### **SAEs**

In addition to reporting all AEs (serious and non-serious) meeting the definitions, the Investigator must report any occurrence of the following as an SAE:

- An ocular infection including a presumed infectious ulcer with any of the following characteristics\*:
  - Central or paracentral location
  - Penetration of Bowman's membrane
  - o Infiltrates > 2 mm diameter
  - Iritis
  - Increase in intraocular pressure
  - Culture positive for microorganisms
  - Increasing size or severity at subsequent visits
- Any central or paracentral corneal event (such as neovascularization) that results in permanent opacification


Status: Effective 

- Hypopyon
- Hyphema
- Neovascularization within the central 6 mm of the cornea
- Permanent vision loss as defined by loss of 2 or more lines of BCVA from enrollment visit that fails to resolve
- Uveitis (anterior, intermediate, or posterior)
- Corneal abrasion affecting  $\geq 50\%$  of corneal surface area

#### Significant Non-Serious AE

A significant non-serious AE is a device-related, non-sight threatening AE that warrants discontinuation of any contact lens wear for greater than or equal to 2 weeks. In addition, the Investigator must report any occurrence of the following as a Significant Non-Serious Adverse Event:

- Peripheral non-progressive non-infectious ulcers
- All symptomatic corneal infiltrative events
- Corneal staining score greater than or equal to Grade 3
- Temporary vision loss as defined by loss of 2 or more lines of BCVA from enrollment visit that persists for 2 or more weeks
- Neovascularization score greater than or equal to Grade 2

# **Device Deficiencies**

A device deficiency is inadequacy of a medical device with respect to its identity, quality, durability, reliability, safety, or performance. A device deficiency may or may not be associated with subject harm (ie, ADE or SADE); however, not all ADEs or SADEs are due


Status: Effective 

to a device deficiency. The Investigator should determine the applicable category listed in the Device Deficiency eCRF for the identified or suspect device deficiency and report any subject harm separately. Examples of device deficiencies include the following:

- Failure to meet product specifications (eg, incorrect lens power/diameter/base curve/color)
- Lens cloudy
- Lens surface/edge defect
- Torn lens during handling/in pack
- Packaging deficit (eg, mislabeled product)
- Suspect product contamination
- Lack of performance

## 11.2 Monitoring for AEs

At each visit, after the subject has had the opportunity to spontaneously mention any problems, the Investigator should inquire about AEs by asking the standard questions:

- "Have you had any health problems since your last study visit?"
- "Have there been any changes in the medicines you take since your last study visit?"



# 11.3 Procedures for Recording and Reporting

AEs are collected from the time of informed consent. Any pre-existing medical conditions or signs/symptoms present in a subject prior to the start of the study (ie, before informed consent is signed) are not considered AEs in the study and should be recorded in the Medical History section of the eCRF.


Status: Effective 

• ADEs or SAEs are documented on the *Serious Adverse Event and Adverse Device Effect* eCRF within 24 hours of the Investigator's or site's awareness.

- Device deficiencies are documented on the *Device Deficiency* eCRF within 24 hours of the Investigator's or site's awareness.
- A printed copy of the completed *Serious Adverse Event and Adverse Device Effect* and/or *Device Deficiency* eCRF must be included with product returns.
- Additional relevant information after initial reporting must be entered into the eCRF as soon as the data become available.
- Document any changes to concomitant medications on the appropriate eCRFs.
- Document all relevant information from Discharge Summary, Autopsy Report,
   Certificate of Death, etc, if applicable, in narrative section of the Serious Adverse
   Event and Adverse Device Effect eCRF.



#### **Intensity and Causality Assessments**

Where appropriate, the Investigator must assess the intensity (severity) of the AE based upon medical judgment with consideration of any subjective symptom(s), as defined below:


Status: Effective 

#### Intensity (Severity)

Mild An AE is mild if the subject is aware of but can easily tolerate the sign or

symptom.

Moderate An AE is moderate if the sign or symptom results in discomfort significant

enough to cause interference with the subject's usual activities.

Severe An AE is severe if the sign or symptom is incapacitating and results in the

subject's inability to work or engage in their usual activities.

For every AE in the study, the Investigator must assess the causality (Related or Not Related to the medical device or study procedure). An assessment of causality will also be performed by Study Sponsor utilizing the same definitions, as shown below:

### Causality

Related An AE classified as related may be either definitely related or possibly related

where a direct cause and effect relationship with the medical device or study procedure has not been demonstrated, but there is a reasonable possibility that

the AE was caused by the medical device or study procedure.

Not Related An AE classified as not related may either be definitely unrelated or simply

unlikely to be related (ie, there are other more likely causes for the AE).



Women of childbearing potential or women who are pregnant at the time of study entry are

Printed By: Print Date:

11.7 Pregnancy in the Clinical Study

not excluded from participation.


Status: Effective 

#### 12 ANALYSIS PLAN

Any deviations to the analysis plan will be updated during the course of the study as part of a protocol amendment or will be detailed in the clinical study report.

All analyses will be conducted according to the applicable statistical analysis plan.

## 12.1 Subject Evaluability

Final subject evaluability must be determined prior to breaking the code for masked treatment (lens) assignment and locking the database, based upon the Deviations and Evaluability Plan.

## 12.2 Analysis Sets

Five analysis sets will be defined:

- a) All Enrolled all subjects signing the informed consent form
- b) Enrolled Dispensed subjects/eyes from All Enrolled that have been exposed to study lenses
- c) Enrolled Not Dispensed subjects/eyes from All Enrolled that have not been exposed to study lenses
- d) Completed Enrolled Dispensed subjects/eyes completing the study
- e) Discontinued Enrolled Dispensed subjects/eyes not complete the study

# 12.3 Demographic and Baseline Characteristics

| Demographic information, | | |
|--------------------------|---|---------------------------------------------|
| | | will be presented by lens group and overall |
| | _ | |

# 12.4 Effectiveness Analyses

For the primary tables will be prepared, when applicable, for the Completed and the Discontinued analysis sets as follows:

- Completed Control (eyes/subjects)
- Completed Test (eyes/subjects)


Status: Effective 

Discontinued Control (eyes/subjects)

• Discontinued Test (eyes/subjects)

No inferential testing will be performed on effectiveness endpoints,

# 12.4.1 Analysis of Primary Effectiveness Endpoint(s)

The primary objective of this study is to demonstrate safety and effectiveness of contact lens when worn for daily wear as compared to Biofinity soft contact lens.

The primary effectiveness endpoint is distance VA with study lenses, collected in Snellen, for each eye. Conversion will be made to the logMAR scale.

# 12.4.1.1 Statistical Hypotheses

No hypothesis testing of the primary effectiveness endpoint is planned.

## 12.4.1.2 Analysis Methods

Alcon - Business Use Only Protocol - Clinical Effective Date: 22-Mar-2019
Status: Effective 

# 12.5 Handling of Missing Data

All data obtained in evaluable subjects/eyes will be used. No imputation for missing values will be carried out.

Incidence and reasons for discontinuation by lens group will be tabulated at each visit and overall.

# 12.6 Safety Analyses

The safety endpoints are:

- AEs
- Biomicroscopy Findings
- Device Deficiencies

There are no safety hypotheses planned in this study. The focus of the safety analysis will be a comprehensive descriptive assessment of occurrence of AE as well as the other listed parameters.

| Alcon - Business Use Only Prot<br>Document: TDOC-0056233<br>Status: Effective | <pre>cocol - Clinical Version: 1.0; CURRENT;</pre> | Effective D<br>Most-Recent; Effective | Page <b>54</b> of <b>59</b> |
|---|---|---|---|
| | nd nargantagas) for a | oular and nanocular A Eq | • |
| Descriptive summaries (counts a | | | |
| presented by Medical Dictionary | • | | <u></u> |
| and Discontinued sets. A listing of | containing details of the | ne AES WIII also de provi | ded. |
| _ | | | |
| 1 | | | |
| 13 DATA HANDLING AN | D ADMINISTRA | TIVE REQUIREM | ENTS |
| 13.1 Subject Confidentiali | ity | | |
| The Investigator must ensure that course of the study. In particular, confidential identifying informat | the Investigator must | keep an enrollment log | with |
| each study participant. | | | |

Alcon - Business Use Only Protocol - Clinical Effective Date: 22-Mar-2019


# 13.2 Completion of Source Documents and Case Report Forms

The nature and location of all source documents will be identified to ensure that original data required to complete the CRFs exist and are accessible for verification by the site monitor, and all discrepancies shall be appropriately documented via the query resolution process. Site monitors are appointed by the Study Sponsor and are independent of study site staff.




Status: Effective 

#### 13.3 Data Review and Clarifications

A review of CRF data to the subject's source data will be completed by the site monitor to ensure completeness and accuracy. After the CRFs have been completed, additional data clarifications and/or additions may be needed as a result of the data cleaning process. Data clarifications are documented and are part of each subject's CRF.

## 13.4 Sponsor and Monitoring Responsibilities

The Study Sponsor will designate a monitor to conduct the appropriate site visits at the appropriate intervals according to the study monitoring plan. The clinical investigation will be monitored to ensure that the rights and well-being of the subjects are protected, the reported data are accurate, complete, and verifiable from the source documents, and the study is conducted in compliance with the current approved protocol (and amendments[s], if applicable), with current GCP, and with applicable regulatory requirements.

The site may not screen subjects or perform the informed consent process on any subject until it receives a notification from an appropriate Study Sponsor representative that the site may commence conducting study activities. Monitoring will be conducted periodically while the clinical study is ongoing. Monitoring methods may include site visits, telephone, written and fax correspondence. Close-out visits will take place after the last visit of the last subject at the site.

A Coordinating Investigator may be identified by the Study Sponsor to review and endorse the final study report. In cases where a Coordinating Investigator is engaged, the Study Sponsor will select the Coordinating Investigator based upon their experience, qualifications, active study participation, and their willingness and availability to take on this role.

# 13.5 Regulatory Documentation and Records Retention

| The Investigator is required to maintain up-to-date, complete regulatory documentation as |
|---|
| indicated by the Study Sponsor and the Investigator's files will be reviewed as part of the |
| ongoing study monitoring. |


Status: Effective 



## 13.6 Quality Assurance and Quality Control

The Study Sponsor will secure agreement from all involved parties to ensure direct access to all study related sites, source data and documents, and reports for the purpose of monitoring and auditing by the Study Sponsor, and inspection by domestic and foreign regulatory authorities. Quality control will be applied to each stage of data handling to ensure that all data are reliable and have been processed correctly. Agreements made by the Study Sponsor with the Investigator/Institution and any other parties involved in the clinical study will be provided in writing as part of the protocol or as a separate agreement.

#### 14 ETHICS



The Investigator must ensure that all personnel involved in the conduct of the study are qualified to perform their assigned responsibilities through relevant education, training, and experience. The Investigator and all clinical study staff must conduct the clinical study in compliance with the protocol. Deviations from this protocol, regulatory requirements and/or GCP must be recorded and reported to the Sponsor prior to database lock. If needed, corrective and preventive action should be identified, implemented, and documented within the study records. Use of waivers to deviate from the clinical protocol is prohibited.

Before clinical study initiation, this protocol, the informed consent form, any other written information given to subjects, and any advertisements planned for subject recruitment must be approved by an IRB/IEC.

Version: 1.0; CURRENT; Most-Recent; Effective **Document:** TDOC-0056233 Status: Effective  Voluntary informed consent must be obtained in writing from every subject and the process shall be documented before any procedure specific to the clinical investigation is applied to the subject. The Investigator must have a defined process for obtaining consent.

Effective Date: 22-Mar-2019

#### 15 REFERENCES

# 15.1 References applicable for all clinical studies

Alcon - Business Use Only Protocol - Clinical

- ISO 11980:2012 Ophthalmic optics Contact lenses and contact lens care products -Guidance for clinical investigations
- ISO 14155:2011 Clinical investigation of medical devices for human subjects Good clinical practice

# 15.1.1 US references applicable for clinical studies

21 CFR Part 11 - Electronic Records; Electronic Signatures


Status: Effective 

• 21 CFR Part 50 - Protection of Human Subjects

- 21 CFR Part 56 Institutional Review Boards
- 21 CFR Part 812 Investigational Device Exemptions
- 21 CFR Part 54 Financial Disclosure by Clinical Investigators
- The California Bill of Rights


Status: Effective